CLINICAL TRIAL: NCT06463249
Title: Scaling up Behavioral Weight Loss Opportunities for Cancer Survivors With Overweight or Obesity in Maryland: A Randomized Trial With Adaptive Interventions (Helpline for Weight Loss)
Brief Title: Behavioral Weight Loss for Cancer Survivors in Maryland: A Trial With Adaptive Interventions
Acronym: Helpline
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Maryland Cigarette Restitution Fund (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00403808
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: All participants will receive Core Helpline intervention in the first two months. If participants achieve 2% or more weight loss in two months (i.e. early responders), they will continue to the Extended Helpline. If participants do not achieve at least 2% of weight loss in two months (i.e. early non-responders), they will be randomized to one of two stepped-up interventions: Enhanced Helpline or Intensive Helpline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intensive Helpline (Experimental): Participants receive 2 scheduled coaching calls/month and individualized coach-scripted feedback via emails twice/month for 6 months.
  Interventions: Behavioral: CORE Helpline; Behavioral: Intensive Helpline
- Enhanced Helpline (Active Comparator): Participants receive 1 participant-initiated call/month. Additionally, the participants receive individualized coach-scripted feedback via emails twice/month for 6 months
  Interventions: Behavioral: CORE Helpline; Behavioral: Enhanced Helpline
- Extended Helpline (Other): Participants who achieved 2% weight loss at 2-month, will continue to Extended Helpline, where the participants can continue receiving 1-on-1 coaching through 1 participant-initiated calls per month for 6 months.
  Interventions: Behavioral: CORE Helpline; Behavioral: Extended Helpline
- CORE Helpline (Other): All participants will receive the CORE Helpline program for 2 months
  Interventions: Behavioral: CORE Helpline

INTERVENTIONS:
Behavioral: CORE Helpline — All participants will receive the Core Helpline program (CORE) for 2 months, which includes written weight loss material, use of a smartphone app, weekly text messages and email reminders and 1 optional participant-initiated coaching call per month.
Behavioral: Extended Helpline — Those who achieved 2% weight loss at 2-month, will continue to Extended Helpline, where the participants can continue receiving all CORE resources including1-on-1 coaching through 1 optional participant-initiated call per month for 6 months.
  Arms: Extended Helpline
Behavioral: Enhanced Helpline — Those who do not reach 2% weight loss at the end of 2 months will be randomized. Participants will continue to receive all CORE resources plus 1 optional participant-initiated call/month for 6 months. Additionally, the participants will receive 2 individualized coach-scripted feedback emails per month, and the option to receive daily text message reminders.
  Arms: Enhanced Helpline
Behavioral: Intensive Helpline — Those who do not reach 2% weight loss at the end of 2 months will be randomized. Participants will continue to receive all CORE resources plus 2 scheduled coaching calls/month for 6 months. Additionally, the participants will receive 2 individual coach-scripted feedback emails per month, and the option to receive daily text message reminders.
  Arms: Intensive Helpline

SUMMARY:
The objective of the HELPLINE Weight Loss Program is to determine the comparative effectiveness of two active multi-component, augmented interventions for cancer survivors with overweight or obesity who do not achieve early weight loss goal in the initial intervention period (termed, early non-responders). The core study design is randomized controlled trial with adaptive intervention.

1. CORE Helpline in all participants (first 2 months)
2. Extended Helpline in early responders (additional 6 months)
3. Enhanced Helpline in early non-responders (additional 6 months)
4. Intensive Helpline in early non-responders (additional 6 months)

DETAILED DESCRIPTION:
All participants will receive

* written Johns Hopkins weight loss material
* instructions for using a smartphone weight loss app to keep track of food and exercise every day (either android or iPhone)
* a weekly weight loss tip by text message and email, and a text message on weight loss progress each week
* a research scale and specific instructions for verifying weights at 5 specific times over the next year.

The participants may also request two 20-minute phone calls during the first 2 months with a weight loss coach.

After the first 2 months, depending on weight loss progress, the participants will be assigned to another program which may include additional assistance for 6 more months.

Additional assistance may include scheduled phone calls with a Johns Hopkins weight loss coach each month, individualized emails from a Johns Hopkins weight loss coach, and the option for daily text message reminders.

After the first 8 months of assistance, the participants will continue the program on the participant's own for 4 more months and provide the study team with final weights 12 months after the start of the program.

ELIGIBILITY:
Inclusion Criteria:

* Women and men ages 18 or older
* Able to complete all study requirements in English
* Have been previously diagnosed with a malignant solid tumor, completed the required surgical, and/or chemotherapy and/or radiation curative intent therapy at least three months prior to enrollment, and have an anticipated treatment-free life span of 12 months or longer. Chemoprophylaxis with tamoxifen or aromatase inhibitors for breast cancer in women and anti- luteinizing hormone-releasing hormone (LHRH) therapy for prostate cancer in men will be permitted.
* Have a BMI ≥ 27 kg/m2 (BMI ≥ 25 kg/m2 for Asians) and weight ≤ 400 lbs.
* Have an email address for regular personal use
* Have a smartphone for personal use, and are willing to use the phone to read emails and text messages, and use an app
* Have adequate data plan and cell service to support daily use of weight loss app, receive text messages and to support coaching calls
* Are willing to record weekly weights
* Are willing to use a tracking app to log food and exercise daily
* Are willing to complete coaching calls as planned
* Are willing to prioritize weight loss efforts by making dietary changes and increasing physical activity

Exclusion Criteria:

* Received any chemotherapy (unless anti-hormonal therapy) and/or radiation three months or less prior to the proposed program date
* Women who are breastfeeding, pregnant, or planning pregnancy within the next year
* self-identification of uncontrolled concurrent medical condition likely to limit compliance with the program as determined by investigators.
* current involvement in another organized weight loss program
* current use of medications known to substantially affect body weight, including chronic oral steroids, Tirzepatide (Mounjaro™), and weight loss doses of other glucagon-like peptide 1 (GLP-1) agonists (e.g. Wegovy.)
* bariatric surgery scheduled within the next 12 months
* plan to move outside the continental United States in the next 12 months
* Weight loss or gain of >5.0% of body weight during 2 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Weight (pounds) changes at 8 months from 2-month between Enhanced Helpline and Intensive Helpline arms | 8 months
  Weight change for Enhanced Helpline and Intensive Helpline in early non-responders

SECONDARY OUTCOMES:
Weight (pounds) change at 5 and 12 months from 2-month between Enhanced Helpline and Intensive Helpline arms | 12 months
  Weight change for Enhanced Helpline and Intensive Helpline in early non-responders

OTHER OUTCOMES:
Weight (pounds) change from baseline to 2 months in all participants | 2 months
  Weight change for CORE Helpline over the first 2 months in all participants
Within-program weight (pounds) changes from baseline to 5, 8, and 12 months in all programs | 12 months
  Weight change for each program over 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Yeh, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins ProHealth, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No